CLINICAL TRIAL: NCT01511874
Title: Non-comparative, Opened Multicenter Study to Assess the Efficacy and Safety of ELIGARD 22.5mg in the Treatment of Subjects With Prostate Cancer
Brief Title: Efficacy and Safety Study of ELIGARD 22.5mg With Prostate Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HanAll BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fr-HE530-01
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Prostate Cancer
Keywords: ELIGARD; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — luprolide acetate gel depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ELIGRAD 22.5mg (Experimental): a subcutaneous injection of ELIGARD 22.5mg at 0 and 12weeks
  Interventions: Drug: ELIGARD 22.5mg

INTERVENTIONS:
Drug: ELIGARD 22.5mg — a subcutaneous injection of ELIGARD 22.5mg at 0 and 12weeks
  Other Names: ELIGARD

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of ELIGARD 22.5mg in the treatment of subjects with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male of 20 years or above
* Subject with prostate cancer with TNM stage T2~4NxMx
* Blood testosterone concentration ≥ 100ng/dl
* Bilirubin ≤ 1.5xULN, transaminase ≤ 2.5xULN
* WHO ECOG performance status ≤ 2
* Signed written informed consent

Exclusion Criteria:

* Hormone-Refractory Prostate cancer
* Brain metastasis
* Another primary malignant tumor except for prostate cancer
* Other conditions which in the opinion of the investigator preclude enrollment into the study

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Ratio of subjects whose blood testosterone concentration is maintained below 50ng/dl at 4 weeks after injection of ELIGARD 22.5mg | 4weeks

SECONDARY OUTCOMES:
Ratio of subjects whose blood testosterone concentration is maintained below 50ng/dL until 24weeks | 24weeks
Ratio of subjects whose blood testosterone concentration exceed 50ng/dL until 24weeks | 24weeks
Change in self assessment scale grade | 0,4, 8, 12, 24 weeks
Ratio of subjects whose blood testosterone concentration is below 20ng/dL at 4weeks and 24weeks | 4, 24 weeks
Change in ECOG performance status | 0,4,8,12, 24weeks
Change in blood prostate-specific antigen | 0,4,8,12,24 weeks
Change in QoL_EPIC grade | 0,12, 24weeks
Change in penile length | screening, 12, 24weeks
Change in testicular volume | screening, 12, 24weeks

CONTACTS AND LOCATIONS:
Overall Officials: Byung Ha Chung, Medicine, Principal Investigator — Department of Urology,Yonsei University,College of Medicine, Gangnam Severance Hospital
Locations (1):
- Department of Urology,Yonsei University,College of Medicine, Gangnam Severance Hospital, Seoul, South Korea